CLINICAL TRIAL: NCT00314925
Title: Phase I Dose-Escalation Study of Seneca Valley Virus (SVV-001), a Replication-Competent Picornavirus, in Patients With Advanced Solid Tumors With Neuroendocrine Features
Brief Title: Safety Study of Seneca Valley Virus in Patients With Solid Tumors With Neuroendocrine Features
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neotropix (Industry)
Responsible Party: Margaret Valnoski, President, Theradex, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N05-10564
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Carcinoid; Neuroendocrine
Keywords: advanced carcinoma; carcinoid; neuroendocrine features; oncolytic virus; phase I study; dose escalation study; rhabdomyosarcoma; alveolar rhabdomyosarcoma; medulloblastoma; rhabdoid; glioblastoma; ewing's sarcoma; pediatric oncologies; neuroblastoma; wilms' tumor; retinoblastoma; Large cell lung cancer
MeSH Terms: conditions — Carcinoid Tumor; Rhabdomyosarcoma; Rhabdomyosarcoma, Alveolar; Medulloblastoma; Glioblastoma; Sarcoma, Ewing; Neuroblastoma; Wilms Tumor; Retinoblastoma | interventions — Biological Factors

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Seneca Valley Virus (biological agent)

INTERVENTIONS:
Drug: Seneca Valley Virus (biological agent) — Dose escalation (starting at 1 × 10^7 vp/kg), IV (in the vein) over 1 hour in a single administration
  Other Names: SVV-001

SUMMARY:
The primary purpose of the study is to determine if Seneca Valley Virus may be administered safely to patients with certain types of advanced cancer.

DETAILED DESCRIPTION:
This is the first study in man of Seneca Valley Virus, a virus which seeks and kills certain tumors in non-human model systems. Subjects in this trial will be patients with advanced cancer displaying certain specified neuroendocrine features, pathologically; they will have exhausted standard methods of treatment for their tumor. The primary purpose of the trial is to determine if the virus may be administered safely. Additional purposes are to learn about the distribution of the virus in the body, the elimination of the virus from the body, the immune response to the virus and whether the virus might have some beneficial effects upon the tumors which the patients have. The first patients will be treated with low amounts of virus and subsequent patients may receive higher amounts. At the end of the trial, it is intended to select a dose for further study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed solid tumor (including carcinoid) with neuroendocrine features (i.e., expression of >= 1 of the following 3 markers: synaptophysin, chromogranin A, or CD56) that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Patients must show evidence of disease progression in the three months prior to treatment with SVV-001.
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of SVV-001 in patients <18 years of age, children are excluded from this study. Children may be eligible for future pediatric Phase I single-agent trials.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Life expectancy >= 24 weeks.
* Adequate bone marrow, hepatic, and renal function as defined below:

  * absolute lymphocyte count >= 1,000/ul
  * absolute neutrophil count >= 1,500/ul
  * platelets >= 100,000/ul
  * AST/ALT <= 2.5 x upper limit of normal (ULN) or <= 5 x ULN if liver metastases present
  * total bilirubin <= 1.5 x upper limit of normal
  * creatinine <= 1.5 x upper limit of normal OR

    * creatinine clearance (calculated) <= 60 mL/min/1.73 m2 for patients with creatinine > 1.5 x upper limit of normal.
* Women must have been surgically sterilized or be post-menopausal.
* Men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for up to 6 months.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients must have oxygen saturation of at least 95% on room air.
* Patients must have measurable disease by RECIST (CT and/or MRI).

Exclusion Criteria:

* Patients with small cell histology.
* Patients who have been hospitalized for emergent conditions requiring inpatient evaluation, treatment or procedure during the 30 days prior to entry on study. In addition, emergent conditions requiring inpatient evaluation, treatment or procedure must have resolved or be medically stable and not severe for 30 days prior to entry on study.
* Use of chemotherapy or radiotherapy within 4 weeks of initiation of SVV-001, or continued > Grade 1 adverse events, excluding alopecia, due to agents administered more than 4 weeks earlier.
* Patients with clinically evident Human Immuno-deficiency Virus (HIV), Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection.
* Patients with > Grade 1 peripheral neuropathy (CTCAE version 3.0).
* Concurrent use of any other investigational agents.
* Presence of or history of central nervous system metastasis.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pre-menopausal women who have not been surgically sterilized. Although SVV-001 has no affect on the ovaries from a toxicological perspective, SVV-001 RNA is present in the ovaries at 12 weeks in animals that were administered high and medium doses. No pre-clinical reproductive tests have been conducted with SVV-001.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity and determination of phase II dose | Within 28 days of treatment administration

SECONDARY OUTCOMES:
Number of responses according to RECIST criteria | Baseline; at Week 7, Day 7 following therapy and then confirmation scan at least 4 weeks later, if required; and every 2 months for up to 6 months, if required
Limited pharmacokinetics, biodistribution and elimination | Until 2 consecutive negative viral assays
Limited evaluation of occurrence of neutralizing antibody | Baseline and at Week 2, Day 1 following therapy

CONTACTS AND LOCATIONS:
Overall Officials: Rudin Charles, MD, PhD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (10):
- United States (10):
  - Cancer Centers of Florida, Ocoee, Florida
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - New York Oncology Hematology P.C., Albany, New York
  - Dayton Oncology & Hematology, P.A ., Kettering, Ohio
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Mary Crowley Research Center, Dallas, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer Specialists - Vancouver Cancer Center, Vancouver, Washington

REFERENCES:
- [Derived] Venkataraman S, Reddy SP, Loo J, Idamakanti N, Hallenbeck PL, Reddy VS. Crystallization and preliminary X-ray diffraction studies of Seneca Valley virus-001, a new member of the Picornaviridae family. Acta Crystallogr Sect F Struct Biol Cryst Commun. 2008 Apr 1;64(Pt 4):293-6. doi: 10.1107/S1744309108006921. Epub 2008 Mar 21. PMID 18391430
- See also: website of sponsor — http://www.neotropix.com